CLINICAL TRIAL: NCT01797601
Title: Insulinsensitivität Des Menschlichen Zentralnervensystems: Kernspintomographische Untersuchung Mit Intranasaler Gabe Von Insulin
Brief Title: Insulin Sensitivity of the Human CNS System: fMRI Study With Intranasal Insulin Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, andreas fritsche, Prof. Andreas Fritsche, University Hospital Tuebingen
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Eudra-CT: 2006-002244-29; 17/2008AMG1 (Other: Ethik-Kommission an der Medizinischen Fakultät der Eberhard-Karls-Universität und am Universitätsklinikum Tübingen)
Record Dates: First submitted 2013-02-18; First posted 2013-02-22 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Obesity; Diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Human Insulin (Active Comparator): Nasal spray
  Interventions: Drug: Human Insulin
- Placebo solution (Placebo Comparator): Nasal spray
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Human Insulin — 160 U of insulin
  Arms: Human Insulin
Drug: Placebo — Insulin dilution medium without insulin
  Arms: Placebo solution

SUMMARY:
The purpose of the study is to investigate whether insulin sensitivity and insulin resistance of the human brain is comparable in all insulin sensitive parts of the brain and whether correlates to other phenotypic information (i.e. whole body insulin sensitivity, BMI, age) of the study participants.

ELIGIBILITY:
Inclusion Criteria:

* Normal routine blood works
* for women: negative pregnancy test
* healthy

Exclusion Criteria:

* Type 2 diabetes
* pregnancy
* acute or chronic diseases
* Pacemakers
* Artificial heart valves
* Metal prostheses
* Implanted magnetic metal parts (screws, ...)
* Metal fragments
* Braces
* insulin pumps
* Tattoos
* claustrophobia
* reduced temperature sensation and / or increased sensitivity to warming of the body
* Ear disease or an increased sensitivity to loud noises

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2013-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Insulin effect on regional brain activity assessed by fMRI | Change from Baseline to 15 minutes and 60 minutes post spray application

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Fritsche, MD, Principal Investigator — Universität Tübingen
Locations (1):
- University of Tuebingen, Tübingen, Germany

REFERENCES:
- [Derived] Kullmann S, Heni M, Veit R, Scheffler K, Machann J, Haring HU, Fritsche A, Preissl H. Selective insulin resistance in homeostatic and cognitive control brain areas in overweight and obese adults. Diabetes Care. 2015 Jun;38(6):1044-50. doi: 10.2337/dc14-2319. Epub 2015 Mar 20. PMID 25795413